CLINICAL TRIAL: NCT01391884
Title: Elimination and Biodegradation of the Incretin Hormones GLP-1 and GIP in Patients With End-stage Renal Disease
Brief Title: Elimination of Incretin Hormones in Patients With Severe Kidney Failure
Status: Completed | Type: Observational
Sponsor: Bo Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, MD DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-2-2009-158-UREMINC
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Uremia
Keywords: Incretin hormones; GLP-1; GIP; Uremia; Dialysis
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dialysis, Non-diabetic: Hemodialysis
- Healthy control

SUMMARY:
The prevalence of type 2 diabetes (T2D) is increasing rapidly worldwide. T2D is characterized by a severely impaired incretin effect. The incretin effect refers to the insulinotropic action of the nutrient-released incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic peptide (GIP). The incretin effect is defined as the difference in insulin secretory responses between oral and isoglycaemic intravenous glucose challenges (OGTT and IIGI, respectively) and in healthy individuals it accounts for as much as 70% of the insulin response following oral glucose, whereas patients with T2D exhibit an incretin effect in the range of 0 to 30%. Patients with T2D and non-diabetic patients with severe kidney failure share several pathophysiological characteristics, including decreased insulin sensitivity, fasting hyperinsulinaemia and impaired beta-cell function. The reason for these findings remains to be fully elucidated. An ongoing study in our research group is investigating the incretin effect and the incretin hormone secretory responses following OGTT, IIGI and meal ingestion, respectively. In continuation of this study, essential knowledge of metabolism of incretin hormones in an uremic milieu will be obtained in the present study prior to evaluation of the use of incretin-based agents in patients with impaired kidney function. In this second study we evaluate the elimination and biodegradation of GLP-1 and GIP. The biological active incretin hormones are rapidly degraded by the ubiquitous enzyme dipeptidyl peptidase-4 (DPP-4), generating inactive metabolites. The active hormones are however also eliminated by renal clearance, although the importance of this remains questionable. It is likely that the degradation and elimination of the active hormones will be significantly affected in patients with severe kidney impairment.

We hypothesize that elimination and biodegradation of the two incretin hormones, both in it´s active and inactive forms, will be affected in non-diabetic patients with severe kidney failure.

ELIGIBILITY:
1)

Inclusion Criteria:

* Male or female; aged 18-90 years
* CKD stage 5 in chronic maintenance dialysis treatment
* BMI: 18,5-28 kg/m2
* Normal fasting plasma glucose (<6,1 mM)
* Normal or impaired glucose tolerance (PG120 min <11,1 mM following OGTT)

Inclusion Criteria:

* Male or female; aged 18-90 years
* Healthy including normal kidney function
* BMI: 18,5-28 kg/m2
* Normal fasting plasma glucose (<6,1 mM)
* Normal or impaired glucose tolerance (PG120 min <11,1 mM following OGTT)

1+2)

Exclusion Criteria:

* Diabetes mellitus
* Chronic pancreatitis / previous acute pancreatitis
* Treatment with oral glucocorticoids, calcineurin inhibitors, thiazides, dipeptidyl peptidase 4 (DPP4) inhibitors or other drugs, which could interfere with glucose or lipid metabolism
* Inflammatory bowel disease
* Malignant disease
* Bowel resection
* Severe anemia (hemoglobin <6.5 mmol/L)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Hemodialysis patients
  2. Healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Intact GLP-1 concentration | -60 min - 180 min
  During GLP-1 infusion 0-60 min
Total GLP-1 concentration | -60 min - 180 min
  GLP-1 infusion 0-60 min
Intact GIP concentration | - 60 min - 180 min
  GIP infusion 0-60 min
Total GIP infusion | -60 min - 180 min
  GIP infusion 0-60 min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology P, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Idorn T, Knop FK, Jorgensen MB, Christensen M, Holst JJ, Hornum M, Feldt-Rasmussen B. Elimination and degradation of glucagon-like peptide-1 and glucose-dependent insulinotropic polypeptide in patients with end-stage renal disease. J Clin Endocrinol Metab. 2014 Jul;99(7):2457-66. doi: 10.1210/jc.2013-3809. Epub 2014 Apr 8. PMID 24712563